CLINICAL TRIAL: NCT07258225
Title: Clinical Effectiveness of a Once-daily Regimen of Tigecycline Compared to the Standard Regimen in Critically Ill Patients
Brief Title: Clinical Effectiveness of a Once-daily Regimen of Tigecycline Compared to the Standard Regimen
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Air Force Specialized Hospital, Cairo, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1.2025
Record Dates: First submitted 2025-11-13; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Multi Drug Resistant Infections
Keywords: Once daily tigecycline; High dose tigecycline; Tigecycline safety; Tigecycline efficacy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm : Usual doses of tigecycline (Active Comparator): Tigecycline standard dose (100 mg loading dose then 50 mg every 12 hours) or (200 mg loading dose then 100 mg every 12 hours). For hepatic patients with a Child-Pugh score (C), the loading dose is 100 mg, then 25 mg every 12 hours
  Interventions: Drug: Usual doses of tigecycline
- Tigecycline once daily regimen (Experimental): Tigecycline once-daily regimen (100 mg once daily) or (200 mg once daily). For hepatic patients with Child-Pugh score (C), the loading dose is 100 mg then 50 mg every 24 hours.
  Interventions: Drug: Tigecycline once daily regimen

INTERVENTIONS:
Drug: Tigecycline once daily regimen — Tigecycline once-daily regimen (100 mg once daily) or (200 mg once daily). For hepatic patients with a Child-Pugh score (C), the loading dose is 100 mg, then 50 mg every 24 hours.
  Arms: Tigecycline once daily regimen
Drug: Usual doses of tigecycline — Tigecycline standard dose (100 mg loading dose then 50 mg every 12 hours) or (200 mg loading dose then 100 mg every 12 hours). For hepatic patients with Child-Pugh score (C), the loading dose is 100 mg then 25 mg every 12 hours
  Arms: Control arm : Usual doses of tigecycline

SUMMARY:
To compare the clinical response (efficacy) and the safety of the tigecycline once daily regimen versus the standard regimen (twice daily regimen). Clinical response was categorized as a cure, failure of treatment, or indeterminate outcome.24 Treatment success (Cure): defined as resolution of signs/symptoms of infection, microbiological cure (negative cultures after tigecycline use), improvement of infection markers (leukocytic count, C reactive protein, and procalcitonin).

Treatment failure: defined as persistence of signs/symptoms of infection despite antimicrobial therapy, deterioration of infection markers (leukocytic count, C reactive protein, and Procalcitonin).

Indeterminate response: subjects who do not have an outcome determination for reasons unrelated to the study drug or infection (e.g., loss to follow-up, withdrawal of consent, etc.) Safety will be assessed by the incidence of adverse events especially which leads to treatment discontinuation.36

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Both males and females.
* Diagnosis of infection has been established and tigecycline use is indicated (intra-abdominal, community-acquired pneumonia, skin Infections) or based on genetic testing and microbiological cultures (MDR Acinetobacter, MDR Stenotrophomonas, MDR Enterobacteriaceae, etc.)

Exclusion Criteria:

* Pregnancy and lactation.
* Bloodstream infections (BSI) and urinary tract infections (UTIs).
* Refusal of attending staff or patient, or family.
* Contraindications to tigecycline, such as hypersensitivity and allergy.
* Patients receiving ≤ 1 day of tigecycline (insufficient length of therapy).
* Patients who have acute physiology and chronic health evaluation (APACHE 2) score of more than 35 (high risk of mortality).
* Do not resuscitate/do not intubate (DNR, DNI) patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Compare treatment outcomes (clinical response) of the tigecycline once-daily regimen and the standard regimen (twice-daily regimen). composite endpoint | 28 days
  Composite clinical response, defined as improvement of inflammatory markers (CRP, Procalcitonin), clinical improvement permitting ICU discharge, and absence of need to modify tigecycline therapy (no escalation or addition of other antibiotics), will be assessed at different time points during the study period. The response is classified as 1- Treatment success (Cure) by improvement of the SOFA score, improvement of infection markers ( CRP, Procalcitonin), and by the need for ICU stay ( ICU length of stay) 2- Treatment failure by an increase of SOFA score, an increase of infection markers ( CRP, Procalcitonin), need to change tigecycline to another antibiotic, or to add on another antibiotic, and death 3) Indeterminate response for drop-out patients and incomplete minimal duration of therapy
Compare the safety of the tigecycline once-daily regimen and the standard regimen (twice-daily regimen). | 28 days
  1. Tigecycline-induced hyperbilirubinemia will be assessed by comparing the baseline bilirubin level to the follow-up level at determined intervals (3 days, 5 days), allowing for comparison of the incidence of hyperbilirubinemia between the two study groups.
  .

SECONDARY OUTCOMES:
- Intensive care unit (ICU) and in-hospital mortality between the two groups. | 28 days
  Calculate the percentage of dead patients in the two groups
Infection markers change between the two groups (C-reactive protein (CRP) | 28 days
  Comparing the increase or decrease in CRP level (mg/L)
Vasopressor needs (only in septic shock patients). | 28 days
  Comparing the duration of vasopressor need between the two groups
Compare the incidence of tigecycline-induced vomiting between the two groups | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Air force specialized hospital, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided